CLINICAL TRIAL: NCT06135025
Title: Evaluation of the Usefulness and Efficacy of Telemonitoring of Patients With COPD
Brief Title: Usefulness and Efficacy of Telemonitoring of Patients With COPD
Acronym: TLM_COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TLM_COPD
Record Dates: First submitted 2023-08-18; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: COPD
Keywords: exacerbation; hospitalization; telemonitoring; acute
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial. Potentially eligible participants are identified using available records from the emergency department of Fattouma Bourguiba Monastir Hospital.
Who Masked: Outcomes Assessor
Masking Description: the outcome assessor was blinded to allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLM_group (Active Comparator): the patients included receive a weekly phone call from the participating physician to to support self-management improvement, use of inhalation devices, rehabilitation, monitoring of signs/symptoms by treatment management, counseling, motivation, and prevention of exacerbations, early recognition of exacerbation signs and planify access to health care facility. at 1 month a Face to Face visit is planned at the pneumology clinic which also unifies the criteria for monitoring and treatment of respiratory disease. Whenever patients came to the emergency room (ER), they were evaluated by the Pneumologist in charge, ergo maintaining a similar approach in the assessment of ERs and deciding whether the patient should be admitted or discharged, independently of their group assignment.
  Interventions: Other: Telemonitoring
- STD_group (No Intervention): Patients in this group receive usual monitoring and treatment regimen is left to the discretion of the treating physicians. At inclusion, patients receive a phone call to collect data.at 1 month a Face to Face visit is planned at the pneumology clinic which also unifies the criteria for monitoring and treatment of respiratory disease. Whenever patients came to the emergency room (ER), they were evaluated by the Pneumologist in charge, ergo maintaining a similar approach in the assessment of ERs and deciding whether the patient should be admitted or discharged, independently of their group assignment.

INTERVENTIONS:
Other: Telemonitoring — the patients included receive a weekly phone call from the participating physician to to support self-management improvement, use of inhalation devices, rehabilitation, monitoring of signs/symptoms by treatment management, counseling, motivation, and prevention of exacerbations, early recognition of exacerbation signs and planify access to health care facility. at 1 month a Face to Face visit is planned to collect data.
  Arms: TLM_group

SUMMARY:
A substantial number of people with COPD suffer from exacerbations, which are defined as an acute worsening of respiratory symptoms. To minimize exacerbations, telehealth has emerged as an alternative to improve clinical management, access to health care, and support for self-management. The study objective was to map the evidence of telehealth/telemedicine for the monitoring of adult COPD patients after hospitalization due to an exacerbation.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major public health problem due to its high prevalence along with high morbi-mortality. Indeed, it is the third leading cause of all-cause death worldwide. COPD is marked by the onset of acute exacerbations (AECOP), which accelerate the progression of the disease, the decline in respiratory function resulting in poor quality of life with a worse survival. Therapeutic education of patients concerning treatment compliance and avoidance of exacerbating factors is one of the means of preventing AECOPD. Education sessions usually occur during during consultations and hospitalizations. Face-to-face visits with health professionals can be hindered by severity of COPD, geographic distance and limited access to health care services.

Telemonitoring patients with COPD could improve delivery of health care, reduce exacerbations, improve quality of life, and results in lower rates of hospitalisation. However, it is unclear whether providing telehealth care improves outcomes of patients with COPD.

This trial aimed to assess the usefulness and efficay of telemonitoring patients with AECOP

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old with prior diagnosis of COPD according to GOLD criteria

Exclusion Criteria:

* dementia
* pregnancy
* reluctance or self-declared inability to engage in the study
* simultaneous participation in another trial involving a therapeutic or non-therapeutic intervention that will interfere with the primary and secondary endpoints of this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Exacerbation rate | 30 days after inclusion
  rate of COPD exacerbation
Need for hospitalization for AECOP | 30 days after inclusion
  rate of hospitalization for AECOP
Mortality | 30 days after inclusion
  rate of Death from any cause

SECONDARY OUTCOMES:
EFI | 30 days after inclusion
  time with free interval from exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Khaoula Bel Haj Ali, MD, Study Director — CHU Fattouma Bourguiba Monastir, service des urgences
Locations (1):
- Khaoula Bel Haj Ali, Monastir, Tunisia